CLINICAL TRIAL: NCT06488222
Title: Intravesical Gemcitabine and Docetaxel for Low Grade Intermediate Risk Bladder Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UF-GU-010; OCR45548 (Other: University of Florida); IRB202401256 (Other: University of Florida)
Record Dates: First submitted 2024-06-21; First posted 2024-07-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; transurethral resection; gemcitabine; docetaxel
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Docetaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Docetaxel and Gemcitabine (Experimental): All subjects will be treated with docetaxel and gemcitabine in 2 phases (induction and maintenance) following transurethral resection. Docetaxel and gemcitabine will be given weekly for six weeks during induction and will then be given every 30 days until up to 12 months after the start of induction therapy during maintenance.
  Interventions: Drug: Docetaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Docetaxel — Subjects will receive 40 mg docetaxel intravesically.
Drug: Gemcitabine — Subjects will receive 1 mg gemcitabine intravesically.

SUMMARY:
Bladder cancer is the 8th most common cancer in the UF Health Cancer Center catchment area and the 7th most common cancer presenting to UFHealth. Most newly diagnosed cases are stage I bladder cancer, which is defined by having no deep muscle invasion and no evidence of disease beyond the bladder. The current use in BCG (Bacillus Calmette-Guerin) refractory disease and the ongoing evaluation in BCG naïve high-risk disease support evaluation of intravesical gemcitabine and docetaxel in decreasing disease recurrence in intermediate risk stage I bladder cancer.

This study will investigate the efficacy and subject compliance with treatment of low grade intermediate risk bladder cancer with intravesical gemcitabine and docetaxel.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age.
* Low-grade (Ta) Intermediate risk urothelial carcinoma of the bladder (defined as recurrent low-grade Ta, solitary low-grade Ta > 3 cm, multifocal low-grade Ta)
* ECOG Performance Status of 0-2.
* No evidence of upper tract urothelial carcinoma based on CT, MRI, or retrograde pyelograms.
* No urethral involvement based on cystoscopy.
* No visible disease based on cystoscopy within 60 days of study enrollment.
* Neutrophil counts ≥ 1500 cells/mm3
* Subjects with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen [as determined by the treating physician or approved by the PI] may be included.
* Subjects of childbearing potential (SOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for at least 6 months after the last dose of study drug to minimize the risk of pregnancy. Prior to study enrollment, subjects of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy.
* Subjects with partners of child-bearing potential must agree to use physician-approved contraceptive methods (e.g., abstinence, condoms, vasectomy) throughout the study and should avoid conceiving children for 3 months following the last dose of study drug.
* Written informed consent obtained from the subject and the subject agrees to comply with all the study-related procedures.

Exclusion Criteria:

* Subjects who have a history of high-grade urothelial carcinoma of the bladder or upper tracts
* Prior treatment with intravesical BCG
* Pure squamous cell carcinoma or adenocarcinoma
* Any component of neuroendocrine carcinoma
* Anatomic abnormalities that prohibit urethral catheter placement
* Low bladder capacity (determined by the treating Urologist) which prohibits treatment with intravesical therapy.
* Subjects of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 6 months after the last dose of study drug.
* Subjects who are confirmed to be pregnant or breastfeeding.
* History of any other disease, metabolic dysfunction, clinical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of protocol therapy or that might affect the interpretation of the results of the study or that puts the subject at high risk for treatment complications, in the opinion of the treating physician.
* Administration of a vaccine containing live virus within 30 days prior to the first dose of trial treatment. Note: Most flu vaccines are killed viruses, with the exception of the intra-nasal vainer (Flu-Mist) which is an attenuated live virus and therefore prohibited for 30 days prior to first dose.
* Prisoners or subjects who are involuntarily incarcerated, or subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Recurrence free survival | 12 months after start of induction
  Evaluate the recurrence free survival, as measured by cystoscopy

SECONDARY OUTCOMES:
Progression rate | 12 months after start of induction
  Determine the progression rate at 12 months, for tumor grade and stage, based on pathologic assessment of tumors in patients with disease recurrence. Development of the following will be considered progression: high grade disease, ≥ T1 disease, CIS.
Treatment compliance | 12 months after the start of induction
  Determine treatment compliance, as measured by how many planned study treatments were given. This will be measured by documented administration of study treatments in the subject's medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Crispen, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States